CLINICAL TRIAL: NCT03723655
Title: A Long-Term Safety Extension Study of Mavacamten (MYK-461) in Adults With Hypertrophic Cardiomyopathy Who Have Completed the MAVERICK-HCM (MYK-461-006) or EXPLORER-HCM (MYK-461-005) Trials (MAVA-LTE)
Brief Title: A Long-Term Safety Extension Study of Mavacamten in Adults Who Have Completed MAVERICK-HCM or EXPLORER-HCM
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CV027-003
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Hypertrophic Cardiomyopathy; Obstructive Hypertrophic Cardiomyopathy; Non-obstructive Hypertrophic Cardiomyopathy
Keywords: Symptomatic, left ventricular outflow tract gradient
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Site, Care Provider and Patients are blinded to study dose. Sponsor is now unblinded to study dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Active Treatment for participants with base target trough concentration
  Interventions: Drug: mavacamten
- Group 2 (Experimental): Active Treatment for participants with higher target trough concentration
  Interventions: Drug: mavacamten
- Group 3 (Experimental): Active Treatment for participants dose titrated to clinical response
  Interventions: Drug: mavacamten

INTERVENTIONS:
Drug: mavacamten — mavacamten capsules
  Other Names: MYK-461

SUMMARY:
Approximately 30 sites that enrolled participants in the MAVERICK-HCM (MYK-461-006) study in the United States (US) will initiate this study.

Approximately 90 sites that enrolled participants in the EXPLORER-HCM (MYK-461-005) study in the US, Europe, and Israel will initiate this study.

Note: Approximately 30 centers overlap between MAVERICK and EXPLORER.

ELIGIBILITY:
Key Inclusion Criteria:

* Has completed the Parent Study through to the EOS Visit within 90 days of consent. (Participants who are beyond the 90-day window from EOS Visit may be included in this study pending MyoKardia Medical Monitoring approval) Participants who prematurely discontinued from the Parent Study or the MAVA-LTE study may be considered for inclusion.
* Has a body weight greater than 45 kg at the Screening Visit
* Has adequate acoustic windows to enable accurate TTEs.
* Has documented LVEF ≥ 50% by echocardiography core laboratory read of screening TTE at rest.
* Has safety laboratory parameters (chemistry, hematology, coagulation, and urinalysis) within normal limits (according to the central laboratory reference range).
* Female participants must not be pregnant or lactating and, if sexually active, must use one of the following highly effective birth control methods from the Screening Visit through 90 days after the last dose of investigational medicinal product (IMP).

In addition to the above contraceptive requirements for female participants, male partners must also use a contraceptive (eg. barrier, condom, or vasectomy).

Key Exclusion Criteria:

* Has any ECG abnormality considered by the investigator to pose a risk to participant safety (eg. second degree atrioventricular block type II).
* Has a history of syncope or a history of sustained ventricular tachyarrhythmia with exercise between Parent Study EOS Visit and Screening Visit.
* Has a history of resuscitated sudden cardiac arrest or known history of appropriate implantable cardioverter-defibrillator (ICD) discharge for life-threatening ventricular arrhythmia between Parent Study EOS Visit and Screening Visit. (Note: history of anti-tachycardia pacing (ATP) is allowed).• Currently treated with disopyramide or ranolazine (within 14 days prior to Screening) or treatment with disopyramide or ranolazine is planned during the study.
* Has any acute or serious comorbid condition (eg. major infection or hematologic, renal, metabolic, gastrointestinal, or endocrine dysfunction) that, in the judgment of the Investigator, could lead to premature termination of study participation or interfere with the measurement or interpretation of the efficacy and safety assessments in the study.
* History of clinically significant malignant disease that developed since enrollment in the Parent Study.
* Is unable to comply with the study requirements, including the number of required visits to the clinical site.
* Has participated in a clinical trial in which the participant received any investigational drug (or is currently using an investigational device) within 30 days prior to Screening, or at least 5 times the respective elimination half-life (whichever is longer), except for participation in MAVERICK-HCM or EXPLORER-HCM. Prior participation in a non-interventional observational study is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events and serious adverse events | 252 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (68):
- United States (31):
  - Local Institution - 0045, Scottsdale, Arizona
  - Local Institution - 0058, Los Angeles, California
  - Local Institution - 0066, San Francisco, California
  - Local Institution - 0063, Stanford, California
  - Local Institution - 0043, New Haven, Connecticut
  - Local Institution - 0067, Jacksonville, Florida
  - Local Institution - 0050, Chicago, Illinois
  - Local Institution - 0070, Indianapolis, Indiana
  - Local Institution - 0049, Iowa City, Iowa
  - Local Institution - 0054, Boston, Massachusetts
  - Local Institution - 0051, Ann Arbor, Michigan
  - Local Institution - 0074, Grand Rapids, Michigan
  - Local Institution - 0048, St Louis, Missouri
  - Local Institution - 0060, New York, New York
  - Local Institution - 0056, New York, New York
  - Local Institution - 0071, Charlotte, North Carolina
  - Local Institution - 0047, Durham, North Carolina
  - Local Institution - 0052, Cincinnati, Ohio
  - Local Institution - 0044, Portland, Oregon
  - Local Institution - 0068, Bethlehem, Pennsylvania
  - Local Institution - 0046, Philadelphia, Pennsylvania
  - Local Institution - 0064, Pittsburgh, Pennsylvania
  - Local Institution - 0073, Memphis, Tennessee
  - Local Institution - 0061, Dallas, Texas
  - Local Institution - 0055, Houston, Texas
  - Local Institution - 0057, Houston, Texas
  - Local Institution - 0072, Murray, Utah
  - Local Institution - 0062, Salt Lake City, Utah
  - Local Institution - 0053, Charlottesville, Virginia
  - Local Institution - 0059, Richmond, Virginia
  - Local Institution - 0065, Seattle, Washington
- Belgium (3):
  - Local Institution - 0002, Aalst
  - Local Institution - 0001, Brussels
  - Local Institution - 0003, Edegem
- Czechia (2):
  - Local Institution - 0010, Prague
  - Local Institution - 0009, Prague
- Denmark (3):
  - Local Institution - 0011, Aarhus
  - Local Institution - 0012, Frederiksberg
  - Local Institution - 0013, Odense
- France (4):
  - Local Institution - 0014, Nantes
  - Local Institution - 0017, Paris
  - Local Institution - 0016, Paris
  - Local Institution - 0015, Toulouse
- Germany (4):
  - Local Institution - 0020, Bad Nauheim
  - Local Institution - 0018, Dresden
  - Local Institution - 0019, Göttingen
  - Local Institution - 0021, Heidelberg
- Israel (6):
  - Local Institution - 0027, Jerusalem
  - Local Institution - 0024, Petah Tikva
  - Local Institution - 0022, Ramat Gan
  - Local Institution - 0025, Rehovot
  - Local Institution - 0023, Safed
  - Local Institution - 0026, Tel Aviv
- Local Institution - 0028, Florence, Italy
- Netherlands (2):
  - Local Institution - 0029, Maastricht
  - Local Institution - 0030, Rotterdam
- Poland (4):
  - Local Institution - 0033, Katowice
  - Local Institution - 0034, Krakow
  - Local Institution - 0031, Poznan
  - Local Institution - 0032, Warsaw
- Portugal (2):
  - Local Institution - 0036, Almada
  - Local Institution - 0035, Lisbon
- Spain (5):
  - Local Institution - 0038, A Coruña
  - Local Institution - 0037, El Palmar
  - Local Institution - 0040, Madrid
  - Local Institution - 0039, Majadahonda
  - Local Institution - 0041, Seville
- Local Institution - 0042, London, United Kingdom

REFERENCES:
- [Derived] Rader F, Oreziak A, Choudhury L, Saberi S, Fermin D, Wheeler MT, Abraham TP, Garcia-Pavia P, Zwas DR, Masri A, Owens A, Hegde SM, Seidler T, Fox S, Balaratnam G, Sehnert AJ, Olivotto I. Mavacamten Treatment for Symptomatic Obstructive Hypertrophic Cardiomyopathy: Interim Results From the MAVA-LTE Study, EXPLORER-LTE Cohort. JACC Heart Fail. 2024 Jan;12(1):164-177. doi: 10.1016/j.jchf.2023.09.028. PMID 38176782
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html